CLINICAL TRIAL: NCT01620411
Title: Management of Chronic Pain in Military Patients With Injuries Sustained During Active Duty. Comparison of Spinal Cord Stimulation and Comprehensive Medical Management.
Brief Title: War Wounded, a Comparison of Two Pain Management Approaches
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Site was never activated by sponsor
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tobias Moeller-Bertram, Associate Clinical Professor of Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120565
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Injuries; Pain
Keywords: Active Duty; Comprehensive Medical Management; Spinal Cord Stimulator; Veteran; sustained; military
MeSH Terms: conditions — Wounds and Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive Medical Management (CMM) (Experimental): This arm will receive standard of care treatment for injuries sustained while on active duty. Non-Invasive.
  Interventions: Other: Comprehensive Medical Management
- CMM + Spinal Cord Stimulator (SCS) (Experimental): This arm will combine comprehensive medical management with placement of a spinal cord stimulator.
  Interventions: Procedure: Spinal Cord Stimulator

INTERVENTIONS:
Other: Comprehensive Medical Management — Standard of care for failed back surgery syndrome sustained while on active duty, primarily focused on physical therapy, medication including: opioid analgesics, muscle relaxants, non-opioid analgesics, etc.
  Arms: Comprehensive Medical Management (CMM)
Procedure: Spinal Cord Stimulator — This arm combines comprehensive medical management (as above) with the trial and possible eventual permenant placement of a spinal cord stimulator, a common pain management procedure.
  Arms: CMM + Spinal Cord Stimulator (SCS)

SUMMARY:
This study aims to investigate the relative effectiveness of two different pain management plans for injuries sustained while active duty in the military. One arm of the study has subjects undergo standard comprehensive medical management, while the other adds the placement of a spinal cord stimulator, a common procedure for the alleviation of pain.

DETAILED DESCRIPTION:
This study aims to investigate the relative effectiveness of two different pain management plans for injuries sustained while active duty in the military. One arm of the study has subjects undergo standard comprehensive medical management, while the other adds the placement of a spinal cord stimulator, a common procedure for the alleviation of pain.

This site was never activated for the research by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a veteran or active duty service member injured while on active military duty receiving care for pain related to the injury(ies) in the Department of Defense health care system or through the Department of Veteran's Affairs.
2. Subject is 18 years of age or older.
3. The elapsed time since the active-duty injury leading to chronic pain is not less than 3 months.
4. Subject reports constant or daily episodes of injury-related pain of at least moderate severity, graded 4 or higher on an 11-point NPRS (point estimate by subject and Investigator at time of enrolment based on overall pain or pain at a specific site). Pain may be nociceptive, neuropathic, or mixed. Phantom pain associated with amputation of an extremity or extremities is allowed.
5. Attempts to control pain with commercially available systemic analgesics have not provided adequate relief, in the judgment of the managing physician and subject.
6. Subject is able to localize site(s) of pain. At least one site of daily pain contributing to moderate severity (Inclusion Criterion 4) and intractability (Inclusion Criterion 5) must be in an extremity, or phantom pain at the site of an amputated extremity. If the extremity site of pain is not an amputated limb, then the pain must have a neuropathic component. This site is identified as the site of Target Pain (TP) for efficacy evaluations during the trial.
7. Subject is an acceptable candidate for surgical placement of an indwelling spinal cord stimulation device.
8. Subject is judged an appropriate candidate for treatment using the available techniques and interventions encompassed within the protocol's definition of comprehensive medical management.
9. For the duration of the trial, subject is willing to limit interventions for control of chronic pain to those approved by the Investigator.
10. The subject is judged psychologically appropriate for either treatment intervention, based on the impression of an interviewing psychologist or psychiatrist.
11. Subject provides informed consent.

Exclusion Criteria:

1. Subject experiences phantom pain associated with amputation of both an upper and lower extremity.
2. Subject has headache or visceral truncal pain or other non-musculoskeletal pain as the only pain that results in constant or daily scores of ≥4 on the 11-point NPRS.
3. Subject has spinal disease that would, in the judgment of the investigator, preclude placement of a spinal cord stimulator.
4. Subject has ongoing chronic infection or a medical condition associated with an unacceptably increased risk of infection related to device implantation.
5. Subject has a current diagnosis or history of psychosis, cognitive impairment, hallucinations, or unexplained loss of consciousness, whether or not related to a combat injury that, in the opinion of the investigator, would exclude the patient from participating in the trial.
6. Subject has a cardiac pacemaker.
7. Subject has any significant medical or psychiatric condition that would interfere with the conduct of the study or with the outcome measures.
8. Subject is pregnant or is breast feeding.
9. Subject has participated in any drug or device trial in the past 30 days.
10. Subject has any planned elective or semi-elective surgery during the 6 months of the Primary Treatment Phase, including stump revisions or grafting.
11. Subject has a psychological condition of great enough severity that it would unacceptably increase the medical risks associated with implantation and care of the devices required for the treatment on the CMM + SCS arm, or would likely interfere with the subject's ability to sustain participation in a research study of long duration. Investigators are encouraged to include the medical monitor and the coordinating investigator in discussions about individual candidate subjects who have psychological diagnoses as part of the polytrauma syndrome before enrollment or treatment on this protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06 (Estimated); Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Decreased Pain Ratings | 3 years
  Pain rating using the Numeric Pain Rating Scale (NPRS) over time. The NPRS is assessing the patients pain on a 11-point rating scale from 0 - 10 with 0 being no pain at all and 10 being the worst imaginable pain. The test is self-reported and can also be administered by an interviewer.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Moeller-Bertram, Principal Investigator — UCSD
Locations (1):
- VA Hospital San Diego, La Jolla, California, United States

REFERENCES:
- See also: Location of study — http://www.sandiego.va.gov/
- See also: Primary Investigator Profile — http://www.va.gov/providerinfo/sandiego/detail.asp?providerid=1409